CLINICAL TRIAL: NCT04174937
Title: A Randomized, Placebo-controlled Study of the Tolerability, Safety and Pharmacokinetics of PA in Healthy Volunteers
Brief Title: PA Tolerability, Safety and Pharmacokinetics in Healthy Volunteers
Acronym: PA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scientific Center for Anti-infectious Drugs, Kazakhstan (Industry)
Collaborators: Institute Of Cardiology & Internal Diseases, Kazakhstan (Other Government); Al-Farabi Kazakh National University (KazNU) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PA-001
Record Dates: First submitted 2017-12-07; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Infections, Respiratory
Keywords: Safety; Iodine complex; Pharmacokinetics; Antibiotic potentiator
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potentiator of antibiotics (PA) (Experimental): Potenciator of antibiotics (PA) , albumin complex of tetraiodid was given per os, single and multiple doses for the different periods (but not exceeding 14 days)
  Interventions: Drug: Potentiator of antibiotics (PA)
- Patients taking placebo PA (Placebo Comparator): Placebo without any active pharmaceutical ingredients was given per os dosed for the patients in same periods of time as per experimental group, single and multiple doses for the different periods (but not exceeding 14 days)
  Interventions: Other: Placebo PA

INTERVENTIONS:
Drug: Potentiator of antibiotics (PA) — Intervention is administered to patients in this Arm
  Other Names: Albumin complex of tetraiodide
  Arms: Potentiator of antibiotics (PA)
Other: Placebo PA — Intervention is administered to patients in this Arm
  Arms: Patients taking placebo PA

SUMMARY:
This is a first-in-human (FIH) study to explore the safety, tolerability and pharmacokinetics of PA after oral ascending dose administration to healthy male volunteers.

DETAILED DESCRIPTION:
The first-in-human dose (FHD) trial is a randomized, double-blind, placebo-controlled, dose-escalation trial assessing safety, tolerability and pharmacokinetics (PK) of single and multiple oral doses of PA in healthy male subjects.

The study consists of two stages: single dose administration and multiple dose administration.

The single dose administration stage includes 5 cohorts, multiple dose administration stage includes at least 4 cohorts (groups). Each cohort includes 8 subjects (6 active drugs and 2 placebos). Cohorts intake ascending doses of study drug. The dose of 1st cohort is 1,0 mg/ml, the doses for the following cohorts will be estimated by the Data Monitoring Committee based on pharmacokinetics and safety results of previous group.

For each subject study includes screening period, one baseline period on Day -1, a treatment period (1 day - at single dose stage; 14 days - at multiple dose stage), followed by safety, PK, assessments up to 72-96 hours post dose. Follow-up visits will take place on Day 7 ; 30; 60 (single dose stage) and 30; 60; 90 (multiple dose stage).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years
* Body mass index 16 to 30
* Subjects should be in good physical and mental health based on medical history, clinical examination and laboratory investigations
* Subjects should have signed informed consent prior to screening and the clinical study after they have read and understood the objective, conduct, risks related to the study, and their rights as study participants
* Subjects should have signed informed consent for being tested for HIV
* Subjects should have signed informed consent to be tested for alcoholemia, use of cannabinoids, cocaine, morphine, benzodiazepines, barbiturates and amphetamine

Exclusion Criteria:

* Subjects should not have evidence of any physical and/or mental health issues at screening and/or results of any clinical, laboratory and/or technical procedures at screening outside of the normal range
* Subjects should not be taking any concomitant medication
* Subjects should not have a history of allergies, hypersensitivity or intolerance to iodine or iodide or to medicines containing iodine such as contrast media used for radiologic examinations
* Subjects should not have a history of addiction or abuse of drugs or alcohol
* Subjects should not be in a position of subordination or other dependence on persons involved in the study such as sponsor, investigators, or any other person or institution interested in its results
* Subjects should not be members of the armed forces or prison inmates
* Subjects should not have positive serology for Hepatitis B, Hepatitis C or HIV
* Subjects should not have any apparent functional and/or physical defects which may or interfere with the study or distort results

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — males
Enrollment: 72 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AE) | Adverse event reporting will be performed throughout the trial from the Screening visit until the Final visit (up to 90 days)
  The safety of ascending single and multiple doses of Study Drug in healthy male subjects will be assessed by adverse event and serious adverse event monitoring.

SECONDARY OUTCOMES:
Area under plasma concentration time curve (AUC∞) | Blood collections at the following time points: before drug intake (two points - 1 day and 10 min), and 5 min, 15 min, 30 min, and 1, 1.5; 2; 3; 6; 9; 12; 15; 24; 48 and 72 hours after study drug administration
  AUC∞ characterizes the total concentration of a drug in serum during the entire observation time. AUC0-∞ is area under the сurve concentration of a drug in blood versus time during the entire observation time. It is calculated on the basis of experimental data. It is measured in μg*hours/liter.
Maximum concentration of drug in the blood (Cmax) | Blood collections at the following time points: before drug intake (two points - 1 day and 10 min), and 5 min, 15 min, 30 min, and 1, 1.5; 2; 3; 6; 9; 12; 15; 24; 48 and 72 hours after study drug administration
  Maximum concentration of drug in the blood after its intake. It is measured in μg /liter.
Time to reach maximum drug concentration (Tmax) | Blood collections at the following time points: before drug intake (two points - 1 day and 10 min), and 5 min, 15 min, 30 min, and 1, 1.5; 2; 3; 6; 9; 12; 15; 24; 48 and 72 hours after study drug administration
  The time required to reach maximum concentration of the drug in blood. Determined by measurements. It is measured in hours.
Half-life time (T1/2) | Blood collections at the following time points: 5 min, 15 min, 30 min, and 1, 1.5; 2; 3; 6; 9; 12; 15; 24; 48 and 72 hours after study drug administration
  The interval of time required to eliminate the half of drug dose from blood. It is calculated on the basis of experimental data. It is measured in hours.
Total clearance (СL) | Blood collections at the following time points: before drug intake (two points - 1 day and 10 min), and 5 min, 15 min, 30 min, and 1, 1.5; 2; 3; 6; 9; 12; 15; 24; 48 and 72 hours after study drug administration
  The total clearance is the volume of plasma from which a substance is completely removed per the unit of time. It is calculated on the basis of experimental data. Clearance is measured in liters / hour * kg of body weight.
Mean residence time of drug (MRT) | Blood collections at the following time points: before drug intake (two points - 1 day and 10 min), and 5 min, 15 min, 30 min, and 1, 1.5; 2; 3; 6; 9; 12; 15; 24; 48 and 72 hours after study drug administration
  MRT is the average time of the drug molecules stays in the body. It is calculated on the basis of experimental data. It is measured in hours.
Drug excretion (%) | Urine samples taken during 0-96 h after drug intake
  Drug excretion with urine over specified periods of time. It is calculated on the basis of experimental data. It is defined as a percentage (%) of single dose or of the total drug amount during its multiple use.It is measured in percents (%).
Volume of distribution (Vλz) | Blood collections at the following time points: 5 min, 15 min, 30 min, and 1, 1.5; 2; 3; 6; 9; 12; 15; 24; 48 and 72 hours after study drug administration
  Volume of distribution is the theoretical volume that would be necessary to contain the total amount of an administered drug at the same concentration that it is observed in the blood plasma. Volume of distribution of the drug in blood is calculated base on terminal phase of drug pharmacokinetic curve. Volume of distribution is an apparent volume that would be necessary to contain the total amount of an administered drug at the same concentration that it is observed in the blood plasma. It is evaluated on the basis of experimental data. It is measured in liters / kg.
Drug elimination rate constant (Lambda-z (λz)) | 0-72 hours
  Drug elimination rate constant in the terminal phase of the pharmacokinetic curve. Elimination rate constant characterizes absorption and excretion. It is measured in 1/hours.
Accumulation index (Rac) | Blood sampling at multiple dosing: Day 1-17
  The degree of accumulation of the drug in the blood at multiple-dose administration. It is evaluated on basis experimental data.
Change in thyroid stimulating hormone (TSH) | Screening visit; Single dose intake: Day 1 - before and 12 hours after dose; Day 2; Day 3; Day 60. Multiple dose intake: Day 1 - before and 12 hours after dosing; Days 2;3;5;9;14;17;30;60;90
  TSH stimulates the thyroid gland to synthesize and secrete thyroid hormone. TSH serum measurements are used to detect primary hypo- and hyperthyroidism. The capability of a TSH assay to distinguish between normal and subnormal concentrations is essential for thyroid testing strategy. It is measured in milli international units per liter (mlU/L). Normal range for the study: 0.5-4.8 mlU/L.
Change in total triiodothyronine (TT3) | Screening visit; Single dose intake: Day 1 - before and 12 hours after dose; Day 2; Day 3; Day 60. Multiple dose intake: Day 1 - before and 12 hours after dosing; Days 2;3;5;9;14;17;30;60;90
  Total triiodothyronine measured in serum and used to diagnose thyroid diseases such as hyperthyroidism and T3-thyrotoxicosis. It is measured in nmol/L. Normal range for the study: 0.85-2.62 nmol/L.
Change in free triiodothyronine (FT3) | Screening visit; Single dose intake: Day 1 - before and 12 hours after dose; Day 2; Day 3; Day 60. Multiple dose intake: Day 1 - before and 12 hours after dosing; Days 2;3;5;9;14;17;30;60;90
  The FT3 is not bound to transport proteins in the circulating blood (unbound T3). It is metabolically active. T3 plays an important role in regulating metabolism. The Free T3 test helps determine whether the thyroid is functioning properly. It is to help diagnose hyperthyroidism and monitor the progress of a patient with a thyroid disorder. It is measured in pmol/L. Normal range for the study: 3.5-6.5 pmol/L.
Change in total thyroxine (TT4) | Screening visit; Single dose intake: Day 1 - before and 12 hours after dose; Day 2; Day 3; Day 60. Multiple dose intake: Day 1 - before and 12 hours after dosing; Days 2;3;5;9;14;17;30;60;90
  Total thyroxine is a hormone used to help diagnose hyper- and hypothyroidism. The TT4 test is usually used with a TSH test to help determine whether the thyroid hormone feedback system is functioning properly, and the results help to distinguish between causes of hyper- and hypothyroidism. It is measured in nmol/L. Normal range for the study: 54 -167 nmol/L.
Change in free thyroxine (FT4) | Screening visit; Single dose intake: Day 1 - before and 12 hours after dose; Day 2; Day 3; Day 60. Multiple dose intake: Day 1 - before and 12 hours after dosing; Days 2;3;5;9;14;17;30;60;90
  The FT4 is an unbound fraction of thyroxine. It is not bound to transport proteins, free in the circulation. The free T4 is metabolically active. It is used in combination with TSH for the diagnosis of thyroid disorders and follow-up of patients with thyroid disorders. It is measured in pmol/L. Normal range for the study: 10-22 pmol/L.
Change in anti-thyroglobulin antibody | Screening visit; Single dose intake: Day 1 - before and 12 hours after dose; Day 2; Day 3; Day 60. Multiple dose intake: Day 1 - before and 12 hours after dosing; Days 2;3;5;9;14;17;30;60;90
  Thyroglobulin (Tg) is a glycoprotein found in thyroid follicular cells that plays a critical role in the biosynthesis of key thyroid hormones. The measurement of anti-TG antibody has been shown to be an aid in the diagnosis of thyroid disorders. It is measured in kilo international units per liter (klU/L). Normal range for the study: up to 40 klU/L.
Change in anti-thyroid peroxidase antibody | Screening visit; Single dose intake: Day 1 - before and 12 hours after dose; Day 2; Day 3; Day 60. Multiple dose intake: Day 1 - before and 12 hours after dosing; Days 2;3;5;9;14;17;30;60;90
  Anti-thyroid peroxidase antibody is a protein found in thyroid follicular cells, is a catalyst in the synthesis of key thyroid hormones. Elevated levels of anti-TPO antibody are a risk factor for autoimmune thyroid diseases. It is measured in klU/L. Normal range for the study: up to 35 klU/L.
Change from baseline in thyroid ultrasound | Screening visit; Final visit (Day 60 - at Single dose intake; Day 90 - at Multiple dose intake)
  Thyroid Ultrasound is used to assess the size of the Thyroid gland and to find out if there are nodules or lesions within the gland. Also the test is used to suspect thyroid disease at screening visit to not include volunteer into the trial.
Change from baseline in electrocardiogram (ECG) | Screening visit; before dose (Day -1); Day 1 - after dose (4 hours); Final visit (Day 60). Multiple dose intake: before dose (Day -1); Day 1 and 15 - 4 hours after dose; Final visit (Day 90).
  A 12-lead resting ECG with a 10 second rhythm strip to be recorded, which includes PR, QT, and QTc intervals as well as QRS interval duration. ECG will be interpreted as "normal", "abnormal, not clinically significant", or "abnormal, clinically significant". Findings classified as "abnormal, clinically significant" will be registered as adverse events if evaluated after dosing.
Change in Respiratory Rate | every visit up to 90 days
  Respiratory rate is an essential vital sign and a fundamental element of patient assessment. It is assessed in combination with heart rate, blood pressure, body temperature. It is measured by counting the breaths (number of times the chest moves up and down) for a full minute in relaxed condition. Normal range for the study is 12-20 breaths per minute.
Change in Heart Rate | every visit up to 90 days
  The heart rate is one of the vital signs. It measures the number of times the heart beats per minute. It is measured in relaxed condition by checking the pulse. To calculate the beats per minute, the patient's pulse is counted for 15 seconds and multiplied by four. Normal range for the study is 60-90 beats per minute.
Change in Blood Pressure | every visit up to 90 days
  Blood Pressure is measured with a sphygmomanometer in a resting condition in three hours after study drug intake, before blood sampling. Subjects should abstain from eating, drinking, smoking one hour before measurement. The bladder should have been emptied. Subject should have been sitting quietly for about 5 minutes before the measurement. Tight clothes should have been removed. Measurements should be taken in sitting position so that the arm and back are supported. Blood Pressure is measured in millimeters of mercury (mm Hg). The systolic and diastolic blood pressure is recorded.
Change in Body Temperature | every visit up to 90 days
  Body Temperature is measured with a mercury thermometer in the armpit in a resting condition three hours after study drug intake, before blood sampling.
Symptoms of musculoskeletal system | From baseline till the last visit (daily during hospital stay, every visit in follow-up period - up to 90 days)
  The symptoms are recorded as a score on a scale. If there are no symptoms the result is reported as "Normal" (score=0). If there are any musculoskeletal symptoms the result is reported as "Abnormal". Each symptom will be estimated as "Clinically non-significant" (score=1) or "Clinically significant"(score=2) and described. The relationship of symptoms with the study drug is assessed as:"Definitely related"(score=3); "Probably related"(score=2); "Possibly related"(score=1); "Not related"(score=0). The scores of clinical significance are summarized with the score of the drug relation. The higher scores mean a worse outcome.
Symptoms of cardiovascular system | From baseline till the last visit (daily during hospital stay, every visit in follow-up period - up to 90 days)
  The symptoms are recorded as a score on a scale. If there are no symptoms the result is reported as "Normal" (score=0). If there are any cardiovascular symptoms the result is reported as "Abnormal". Each symptom will be estimated as "Clinically non-significant" (score=1) or "Clinically significant"(score=2) and described. The relationship of symptoms with the study drug is assessed as:"Definitely related"(score=3); "Probably related"(score=2); "Possibly related"(score=1); "Not related"(score=0). The scores of clinical significance are summarized with the score of the drug relation. The higher scores mean a worse outcome.
Symptoms of lymphatic system | From baseline till the last visit (daily during hospital stay, every visit in follow-up period - up to 90 days)
  The symptoms are recorded as a score on a scale. If there are no symptoms the result is reported as "Normal" (score=0). If there are any lymphatic symptoms the result is reported as "Abnormal". Each symptom will be estimated as "Clinically non-significant" (score=1) or "Clinically significant"(score=2) and described. The relationship of symptoms with the study drug is assessed as:"Definitely related"(score=3); "Probably related"(score=2); "Possibly related"(score=1); "Not related"(score=0). The scores of clinical significance are summarized with the score of the drug relation. The higher scores mean a worse outcome.
Symptoms of nervous system | From baseline till the last visit (daily during hospital stay, every visit in follow-up period - up to 90 days)
  The symptoms are recorded as a score on a scale. If there are no symptoms the result is reported as "Normal" (score=0). If there are any nervous symptoms the result is reported as "Abnormal". Each symptom will be estimated as "Clinically non-significant" (score=1) or "Clinically significant"(score=2) and described. The relationship of symptoms with the study drug is assessed as:"Definitely related"(score=3); "Probably related"(score=2); "Possibly related"(score=1); "Not related"(score=0). The scores of clinical significance are summarized with the score of the drug relation. The higher scores mean a worse outcome.
Symptoms of Respiratory system | From baseline till the last visit (daily during hospital stay, every visit in follow-up period - up to 90 days)
  The symptoms are recorded as a score on a scale. If there are no symptoms the result is reported as "Normal" (score=0). If there are any Respiratory symptoms the result is reported as "Abnormal". Each symptom will be estimated as "Clinically non-significant" (score=1) or "Clinically significant"(score=2) and described. The relationship of symptoms with the study drug is assessed as:"Definitely related"(score=3); "Probably related"(score=2); "Possibly related"(score=1); "Not related"(score=0). The scores of clinical significance are summarized with the score of the drug relation. The higher scores mean a worse outcome.
Symptoms of Gastrointestinal system | From baseline till the last visit (daily during hospital stay, every visit in follow-up period - up to 90 days)
  The symptoms are recorded as a score on a scale. If there are no symptoms the result is reported as "Normal" (score=0). If there are any gastrointestinal symptoms the result is reported as "Abnormal". Each symptom will be estimated as "Clinically non-significant" (score=1) or "Clinically significant"(score=2) and described. The relationship of symptoms with the study drug is assessed as:"Definitely related"(score=3); "Probably related"(score=2); "Possibly related"(score=1); "Not related"(score=0). The scores of clinical significance are summarized with the score of the drug relation. The higher scores mean a worse outcome.
Symptoms of urinary system | From baseline till the last visit (daily during hospital stay, every visit in follow-up period - up to 90 days)
  The symptoms are recorded as a score on a scale. If there are no symptoms the result is reported as "Normal" (score=0). If there are any urinary symptoms the result is reported as "Abnormal". Each symptom will be estimated as "Clinically non-significant" (score=1) or "Clinically significant"(score=2) and described. The relationship of symptoms with the study drug is assessed as:"Definitely related"(score=3); "Probably related"(score=2); "Possibly related"(score=1); "Not related"(score=0). The scores of clinical significance are summarized with the score of the drug relation. The higher scores mean a worse outcome.
Symptoms of Endocrine system | From baseline till the last visit (daily during hospital stay, every visit in follow-up period - up to 90 days)
  The symptoms are recorded as a score on a scale. If there are no symptoms the result is reported as "Normal" (score=0). If there are any endocrine system symptoms the result is reported as "Abnormal". Each symptom will be estimated as "Clinically non-significant" (score=1) or "Clinically significant"(score=2) and described. The relationship of symptoms with the study drug is assessed as:"Definitely related"(score=3); "Probably related"(score=2); "Possibly related"(score=1); "Not related"(score=0). The scores of clinical significance are summarized with the score of the drug relation. The higher scores mean a worse outcome.
Symptoms of Skin and subcutaneous tissue | From baseline till the last visit (daily during hospital stay, every visit in follow-up period - up to 90 days)
  The symptoms are recorded as a score on a scale. If there are no symptoms the result is reported as "Normal" (score=0). If there are any skin and subcutaneous tissue symptoms the result is reported as "Abnormal". Each symptom will be estimated as "Clinically non-significant" (score=1) or "Clinically significant"(score=2) and described. The relationship of symptoms with the study drug is assessed as:"Definitely related"(score=3); "Probably related"(score=2); "Possibly related"(score=1); "Not related"(score=0). The scores of clinical significance are summarized with the score of the drug relation. The higher scores mean a worse outcome.
Change in Alanine transaminase (ALT) | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  The ALT test measures the amount of ALT in the blood. High levels of ALT in the blood can indicate a liver problem, even before clinical signs of liver disease. It is measured in IU/L. Normal range for the study: ≤ 45 IU/L.
Change in Aspartate aminotransferase (AST) | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  The AST blood test measures the amount of AST in the blood. AST is an enzyme that is found mostly in the liver. AST releases into bloodstream when liver is damaged. The test can help to diagnose liver damage or disease. It is measured in IU/L. Normal range for the study: ≤ 41 IU/L.
Change in Bilirubin / bilirubin fractions | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  The level of bilirubin is measured in the blood by the bilirubin blood test. Direct bilirubin is water-soluble form of bilirubin. Indirect bilirubin is fat-soluble form of bilirubin.
  Direct and indirect are measured solely. Total and direct bilirubin levels can be measured from the blood, but indirect bilirubin is calculated from the total and direct bilirubin. It is measured in μmol/L. Normal range for the study: 8,6-20,5 μmol/L.
Change in Creatinine | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Serum creatinine is measured in the blood. Creatinine measurements are used in the trial as the indicator of kidney function. Elevated creatinine level signifies impaired kidney function or kidney disease. As the kidneys become impaired for any reason, the creatinine level in the blood will rise due to poor clearance of creatinine by the kidneys. Abnormally high levels of creatinine thus warn of possible malfunction or failure of the kidneys. It is measured in μmol/L. Normal range for the study: ≤133 μmol/L.
Change in Alkaline phosphatase | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  The alkaline phosphatase is measured in the blood. High levels of alkaline phosphatase may indicate the liver damage. It is measured in IU/L. Normal range for the study: 40-129 IU/L.
Change in Blood Urea Nitrogen | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  The amount of urea nitrogen is measured in the blood. The urea is produced by liver in the urea cycle as a waste product of the digestion of proteins. The elevated levels of Blood Urea Nitrogen may be a sign that that kidneys aren't working efficiently. The accumulation of urea and other nitrogen-containing compounds in the blood due to renal failure leads to uremia. The main causes of an increase in Blood Urea Nitrogen are: high protein diet, decrease in glomerular filtration rate (suggestive of renal failure), decrease in blood volume (hypovolemia), congestive heart failure, gastrointestinal hemorrhage,[4] fever, and increased catabolism. Hypothyroidism can cause both decreased glomerular filtration rate and hypovolemia, but Blood Urea Nitrogen -to-creatinine ratio has been found to be lowered in hypothyroidism and raised in hyperthyroidism. It is measured in mmol/L. Normal range for the study: ≤8.3 mmol/L.
Change in Uric acid | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Uric acid is a product of the metabolic breakdown of purine nucleotides, and it is a normal component of urine. High blood concentrations of uric acid may be caused by study drug, hypothyroidism, kidney damage and called hyperuricemia. It can lead to gout and are associated with other medical conditions, including diabetes and the formation of ammonium acid urate kidney stones.
  Uric acid in blood is measured in mmol/L. Normal range for the study: ≤480 mmol/L.
Change in Alpha-amylase (α-amylase) | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  α-amylase is an enzyme that catalyze the hydrolysis of starch into smaller carbohydrate molecules.
  The alpha-amylase is produced by the salivary glands, whereas pancreatic amylase is secreted by the pancreas into the small intestine. Both the salivary and pancreatic amylases are α-amylases.
  Blood serum amylase may be increased in case of the pancreas damage by the study drug. α-amylase in blood is measured in mmol/L. Normal range for the study: 28-100 U/L
Change in Serum total protein | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Protein in the serum consists of albumin and globulin. Protein fractions are determined using electrophoresis. Total protein levels in the blood give a general indication of the state of hydration, nutrition or proper functioning of certain major organs such as the liver, kidneys or bone marrow. Total protein in blood is measured in g/L. Normal range for the study: 64-83 g/L. Concentrations below the reference range may be a sign of low albumin concentration, liver damage, acute inflammation, or a problem of malnutrition or malabsorption of amino acids necessary for protein formation. It may be also a sign of immunodeficiency. Too much protein loss from the kidneys or too much water in the blood can also cause hypoproteinemia. Concentrations above the reference range (hyperproteinemia) may indicate dehydration or an increase in the gammaglobulin fraction, as found in chronic inflammatory diseases, certain viral infections or bone marrow disorders.
Change in Albumin level in blood | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Albumin is a protein made by the liver. Albumin is measured in the blood. Albumin carries substances such as hormones, medicines, and enzymes throughout the body. Low albumin levels can indicate a problem with the liver or kidneys. Albumin in blood is measured in g/L. Normal range for the study: 35-55 g/L.
Change in Glucose level in blood | Single dose study:Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose study: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Measuring blood glucose levels is primarily used to monitor blood sugar levels to diagnose hyperglycemia or hypoglycemia caused by study drug. It is measured in fasting condition. Glucose in blood is measured in mmol/L. Normal range for the study: 4,11-5,89 mmol/L.
Change in Total cholesterol | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  It is measured in the blood. It includes all the cholesterol in all the lipoprotein particles: high-density lipoprotein cholesterol (HDL) and low-density lipoprotein cholesterol (LDL).
  Total cholesterol in blood is measured in mmol/L. Normal range for the study: ≤5.2 mmol/L. It is used to diagnose the metabolism of lipids and the liver function.
Change in Potassium in blood | Single dose study:Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose study: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Measurement of the amount of potassium in the blood helps to diagnose an electrolyte imbalance caused by study drug. Changed potassium level (hypokaliemia, hyperkaliemia) may cause such problems as muscle weakness or contractions, nerve signals transmission, cardiac arrhythmia, hypertension, may affect the kidney function and hormone release. Potassium in the blood is measured in mmol/L. Normal range for the study: 3.5 - 5.3 mmol/L
Change in Serum calcium | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Measurement of the amount of calcium in the blood helps to diagnose an electrolyte imbalance caused by study drug. Changed calcium level (hypocalcaemia, hypercalcaemia) may influence the proper functioning of muscles, nerves, and the heart, coagulation, maintenance of bones and teeth.Calcium in the blood is measured in mmol/L. Normal range for the study: 2,15-2,55 mmol/L.
Change in Serum magnesium | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Measurement of the amount of magnesium in the blood helps to diagnose an electrolyte imbalance caused by study drug. Abnormal levels of magnesium may influence the proper functioning of muscles, nerves, and the heart, helps control blood pressure and blood sugar. Low level of magnesium in the body may cause numerous symptoms: poor coordination, muscle spasms, loss of appetite, personality changes, and nystagmus. Magnesium in the blood is measured in mmol/L. Normal range for the study: 0,65- 1,5 mmol/L.
Change in erythrocytes number in blood | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  The influence of the study drug on the number and morphology of erythrocytes will be assessed. Normal range for the study: 3,9-5,5 х10^12 per liter.
Change in hemoglobin | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  The influence of the study drug on to the amount of hemoglobin will be assessed. Normal range for the study: 130-180 g/L.
Change in leucocytes number in the blood | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  The influence of the study drug on the number and morphology of leucocytes will be assessed. Normal range for the study: 4,0-9,0 х10^9 per liter.
Change in thrombocytes number in the blood | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  The influence of the study drug on the number and morphology of thrombocytes will be assessed. Normal range for the study: 180-400 х10^9 per liter.
Change in hematocrit | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  It is the percentage of red blood cells (RBC's) in the blood. The hematocrit test indicates the percentage of blood by volume that is composed of red blood cells. A hematocrit is measured in L/L (litre of cells per litre of blood). Normal range for the study: 36-55% .
Change in Erythrocyte Sedimentation Rate (ESR)) | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  ESR indirectly measures the degree of inflammation present in the body. The test actually measures the rate sedimentation of erythrocytes in a sample of blood that has been placed into a tall, thin, vertical tube. Results are reported as the millimeters of plasma that are present at the top portion of the tube after one hour. The ESR is non-specific test that provides general information about the presence or absence of an inflammatory condition. Normal range for the study: 2-10 mm/hour.
Change in prothrombin index | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 15;16;17;30;60;90
  Measured in percents. Normal range for the study: 70-130 %
Change in activated partial thromboplastin time (aPTT) | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 15;16;17;30;60;90
  Measured in seconds. Normal range for the study: 23-38 seconds
Change in prothrombin ratio | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 15;16;17;30;60;90
  The ratio of a patient's prothrombin time to a normal (control) sample, raised to the power of the ISI value for the analytical system being used. Measured as a ratio. Normal range for the study:0,9-1,2
Change in thrombin time | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 15;16;17;30;60;90
  Thrombin clotting time measures the time it takes for a clot to form in the plasma of a blood sample containing anticoagulant, after an excess of thrombin has been added.Measured in seconds. Normal range for the study:15-21 seconds
Change of protein level in urine | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Proteinuria caused by study drug will be assessed. It may be due to kidney damage, heart failure, loss of body fluids (dehydration), high blood pressure. Protein level in urine is measured in mg/L.
Change in Urinary glucose | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Glycosuria caused by study drug will be assessed. Measured in mmol/L Normal range for the study: 0 to 0.8 mmol/L.
Hematuria | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Hematuria caused by study drug will be assessed.It is measured in the number of red blood cells per high-power field in microscopic investigation of urine sediment.
Leucocyturia | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Leucocytes in urine after study drug intake will be assessed. Leucocyturia may be due to inflammation of the urinary track or adjacent tissue. It is measured in the number of white blood cells per high-power field in microscopic investigation of urine sediment.
Ketonuria | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  Ketone bodies present in the urine after study drug intake will be assessed. It may be due to excess ketones production as an indication that the body is using an alternative source of energy. It is measured in mg/dL. A negative test result is normal.
  An abnormal result: small ketonuria: <20 mg/dL; moderate ketonuria: 30 to 40 mg/dL; large ketonuria: >80 mg/dL
Change in urine pH | Single dose intake: Screening visit; before dose (Day -1); Day 1 - after dose (3 hours); Days 2;7;30;60. Multiple dose intake: Screening visit; before dose (Day -1); Days 1; 3;10;14-after dose (3 hours); Days 17;30;60;90
  The influence of study drug on to urine pH will be evaluated. The normal values range from pH 4.6 to 8.0
Change in immunoglobulin A (IgA) level in blood | Single dose study: before dose (Day -1); Day 1 - after dose (3 hours); Day 2. Multiple dose study: before dose (Day -1) Days 14; 17; 30;60; 90
  The influence of study drug onto IgA level in blood will be evaluated. It is measured in g/L. Normal range for the study: 0,7-4,0 g/L.
Change in immunoglobulin M (IgM) level in blood | Single dose intake: before dose (Day -1); Day 1 - after dose (3 hours); Day 2. Multiple dose intake: before dose (Day -1) Days 14; 17; 30;60; 90
  The influence of study drug onto IgM level in blood will be evaluated. It is measured in g/L. Normal range for the study: 0,4-2,3 g/L.
Change in immunoglobulin G (IgG) level in blood | Single dose intake: before dose (Day -1); Day 1 - after dose (3 hours); Day 2. Multiple dose intake: before dose (Day -1) Days 14; 17; 30;60; 90
  The influence of study drug onto IgG level in blood will be evaluated. It is measured in g/L. Normal range for the study: 7-16 g/L.
Change in immunoglobulin E (IgE) level in blood | Single dose intake: Screening visit; Day 1 - after dose (3 hours); Day 2. Multiple dose intake: Screening visit; Days 14; 17; 30;60; 90
  The influence of study drug onto IgE level in blood will be evaluated. It is measured in IU/ml . Normal range for the study: 0,100-200,0 IU/ml.
Change in Rheumatoid factor | Single dose intake: Screening visit; Day 1 - after dose (3 hours); Day 2. Multiple dose intake: Screening visit; Days 14; 17; 30;60; 90
  The influence of study drug onto Rheumatoid factor in blood will be evaluated. It is measured in IU/ml . Normal range for the study: 0-25 IU/ml.
Change in C-Reactive Protein | Single dose intake: Screening visit; Day 1 - after dose (3 hours); Day 2. Multiple dose intake: Screening visit; Days 14; 17; 30;60; 90
  The influence of study drug onto C-Reactive Protein in blood will be evaluated. It is measured in mg/l . Normal range for the study: 0-5 mg/l
Change in Antimitochondrial Antibody | Single dose intake: before dose (Day -1); Day 30; Day 60. Multiple dose intake: before dose (Day -1); Day 60; Day90
  The influence of study drug on Antimitochondrial Antibody in blood will be evaluated. It is measured in IU/ml. Normal range for the study: 0-10 IU/ml
Change in antinuclear antibody | Single dose intake: before dose (Day -1); Day 30; Day 60. Multiple dose intake: before dose (Day -1); Day 60; Day90
  The influence of study drug on antinuclear antibody in blood will be evaluated. It is measured in IU/ml. Normal range for the study: 0-40 IU/ml
Change from baseline in CD3+tcells | Single dose intake: before dose (Day -1); Day 1 - after dose (3 hours); Days 2; 17; 30; 60. Multiple dose intake: before dose (Day -1); Day 1; 14 - after dose (3 hours); Days 17;30;60;90
  The influence of study drug on CD3+ tcells percent in blood will be evaluated. Normal range for the study: 52-76 %
Change from baseline in CD4+tcells | Single dose intake: before dose (Day -1); Day 1 - after dose (3 hours); Days 2; 17; 30; 60. Multiple dose intake: before dose (Day -1); Day 1; 14 - after dose (3 hours); Days 17;30;60;90
  The influence of study drug on CD4+ tcells percent in blood will be evaluated. Normal range for the study: 31-46 %
Change from baseline in CD8+tcells | Single dose intake: before dose (Day -1); Day 1 - after dose (3 hours); Days 2; 17; 30; 60. Multiple dose intake: before dose (Day -1); Day 1; 14 - after dose (3 hours); Days 17;30;60;90
  The influence of study drug on CD8+ tcells percent in blood will be evaluated. Normal range for the study: 23-40 %
Change from baseline in Ratio CD4/CD8 | Single dose intake: before dose (Day -1); Day 1 - after dose (3 hours); Days 2; 17; 30; 60. Multiple dose intake: before dose (Day -1); Day 1; 14 - after dose (3 hours); Days 17;30;60;90
  The influence of study drug on Ratio CD4/CD8 in blood will be evaluated. Normal range for the study: 1.2-2.0 %

CONTACTS AND LOCATIONS:
Overall Officials: Amirkan A Azembayev, PhD, Study Director — JSC "Scientific Center for Anti-infectious Drugs"
Locations (1):
- Institute Of Cardiology & Internal Diseases, Almaty, Almatinskaya, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Structure and possible mechanism of action of new drug — https://www.ncbi.nlm.nih.gov/pubmed/22332742
- See also: Interaction of iodine complexes with viral DNA — https://link.springer.com/chapter/10.1007%2F978-1-4899-7699-4_10
- See also: Quantitative Determination of Iodide Ions in Substances and Tablets Containing Iodine Adducts — https://www.rjpbcs.com/pdf/2016_7(6)